CLINICAL TRIAL: NCT05743439
Title: Early Augmentative and Alternative Communication (AAC) Intervention Delivered Via Hybrid Telehealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Florida State University (Other)
Responsible Party: Principal Investigator, Emily Quinn, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021611
Record Dates: First submitted 2023-02-13; First posted 2023-02-24 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Intellectual Disability; Speech and Language Disorder
MeSH Terms: conditions — Intellectual Disability; Speech; Language Disorders | interventions — Methods

STUDY DESIGN:
Masking Description: Although this is a single-arm trial, outcome assessors will be masked to reduce potential for experimenter bias. We will also employ a technique for single-case experimental designs called masked visual analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Augmentative and Alternative Communication (AAC) Intervention (Experimental): After a period of stable baseline performance (3 to 5 sessions) on parent and child outcomes, the interventionist will apply the early AAC intervention.
  Interventions: Behavioral: Early Augmentative and Alternative Communication (AAC) Intervention

INTERVENTIONS:
Behavioral: Early Augmentative and Alternative Communication (AAC) Intervention — Caregivers will receive 24, 50 min intervention sessions twice a week for three months. During each intervention session, the therapist provides instruction and coaching on using AAC and a set of evidence-based language support strategies. Strategies are taught sequentially in three phases: (1) Responding to all Communication, (2) Teaching Words, and (3) Creating Communication Opportunities. Caregivers practice using the AAC intervention strategies during three, five-minute routines with their children. Therapists coach the caregiver on using the targeted strategies during these routines, encouraging caregivers to reflect on their implementation, and developing a plan to use the AAC strategies during activities not practiced during the intervention session. The AAC intervention is provided to families using an evidence-based service delivery model, Family Guided Routines Based Intervention.

SUMMARY:
The goal of this mixed methods study aims to develop and pilot test an augmentative and alternative communication (AAC) intervention for toddlers with intellectual and developmental disabilities (IDD) and their families. The main question it aims to answer is: Will this AAC intervention improve caregivers' use of naturalistic AAC intervention strategies, leading to increases in children's communication? The investigators will employ qualitative methods to conduct interviews to determine caregiver and speech-language pathologist preferences regarding an AAC intervention. Findings from these interviews will inform the adaptation of the AAC intervention procedures, service delivery approach, and strategies to increase caregiver's treatment adherence. Next, the researchers will conduct six multiple baseline designs across behaviors (AAC strategies) to develop the AAC intervention and demonstrate preliminary efficacy when delivered to families in-person. Caregiver-child dyads will receive 24 in-person intervention sessions during which the therapist will provide AAC instruction and coaching on using AAC strategies to caregivers. Last, the investigators will pilot test the AAC intervention using a hybrid telehealth model with nine caregiver-child dyads. Caregiver-child dyads will receive 24 intervention sessions, eight sessions provided to families in-person, and 16 sessions provided to families via telehealth.

Our long-term goal is to develop a socially valid and effective intervention to improve language outcomes for toddlers with IDD. The researchers propose developing and pilot testing a hybrid telehealth AAC intervention for toddlers with IDD and their families. Researchers employ an implementation science approach, using systematic qualitative methods to identify caregivers' preferences and single-case experimental design methods to assess the feasibility of the AAC intervention. The central hypothesis is that the intervention will improve caregivers' use of naturalistic AAC intervention strategies, leading to increases in children's communication.

DETAILED DESCRIPTION:
Aim 1: Determine stakeholders' preferences and needs for two key AAC intervention components: (a) service delivery and (b) strategies to enhance treatment adherence. Researchers will conduct and analyze interviews with ten caregivers and ten speech-language pathologists (SLPs) to assess the acceptability of different service delivery models (e.g., in person, telehealth, hybrid). Interviews will also focus on identifying strategies (e.g., text-message reminders, video modeling) with the potential to support caregivers' adherence and promote generalization to new activities. Results will inform AAC intervention development (Aim 2).

Aim 2: Develop an AAC intervention through iterative testing cycles. Researchers will conduct six multiple-baseline designs to investigate the effects of an AAC intervention on caregivers' AAC intervention strategy use (primary outcome) and children's communication acts (secondary outcome). Six caregiver-child dyads will receive 24 in-person intervention sessions, during which the therapist will teach caregivers to use AAC and language facilitation strategies during family-selected routines. Social validity will be assessed via weekly questionnaires and a post-intervention interview. In this experiment, the feasibility of in-person delivery is investigated to establish the acceptability and effects of the intervention procedures before pilot testing hybrid delivery. Results will inform modifications which will be tested in a hybrid delivery model (Aim 3).

Aim 3: Conduct a pilot test of a hybrid telehealth AAC intervention. Researchers will employ a combination multiple probe design to investigate the feasibility of a hybrid telehealth AAC intervention. Nine caregiver-child dyads will receive 24 intervention sessions (8 in-person, 16 telehealth) which include coaching on AAC and language facilitation strategies. The investigators hypothesize that the intervention will increase caregivers' AAC intervention strategy use (primary outcome) and children's communication acts (secondary outcome). Child communication outcomes and caregivers' social validity assessments will be explored to inform a future large-scale trial.

ELIGIBILITY:
1. Speech-Language Pathologists:

   1. age > 18 years
   2. full or part-time employment providing language intervention to children 24 - 36 months with IDD
   3. has at least 1 child on their caseload who uses AAC
   4. has 2 or more years of experience providing AAC to children with IDD
   5. able to speak, understand, and read English.
2. Caregivers:

   1. age > 18 years
   2. parent, primary caregiver, or legal guardian of a child age 24 - 36 months with IDD
   3. has at least 6 months of experience receiving early intervention, and
   4. able to speak, understand, and read English.
3. Children:

   1. age 24 - 36 months
   2. diagnosis of IDD confirmed by caregiver or medical record
   3. severe developmental delay, defined as a score of > 2 standard deviations below the mean on the Mullen Scales of Early Learning (MSEL) Early Learning Composite
   4. severe expressive language impairment, defined as a score of < 12 months on the Expressive Language Subscale of the MSEL and expressive vocabulary and < 10 words (signs, or symbols) per caregiver report on the MacArthur-Bates Communicative Development Inventories Words and Gestures (MCDI-WG)
   5. receptive vocabulary of at least 50 words, per caregiver report on MCDI-WG
   6. use of intentional communication behaviors, defined as a score of > 7 on the Communication Complexity Scale
   7. sufficient motor skills to sit upright with support, interact with toys provided during the assessment, and access the AAC system
   8. hearing within normal limits, defined as 0 to 25 dbHL in at least one ear
   9. vision within normal limits, defined as 20/80 visual acuity or better in at least one eye, and
   10. exposure to English in the home or community.
   11. Children with uncontrolled seizure disorders will be excluded.

Min Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Caregiver Use of AAC Intervention Strategies | Assessed 1-2 times per week through study completion, 3-4 months.
  Observational assessment of caregivers' use of AAC strategies during a 15-min caregiver-child interaction. The primary dependent variable is the caregiver's use of AAC strategies. The metric is the accuracy of AAC strategy use calculated by (correct strategy steps/ total strategy steps X100).

SECONDARY OUTCOMES:
Change in Number of Child Communication Acts | Assessed 1-2 times per week through study completion, 3-4 months.
  Observational measure of a child's expressive communication behaviors including gestures, vocalizations, spoken words, manual signs, and picture symbols during a 15-min caregiver-child interaction. The secondary dependent variable is the number of child communication acts expressed. The metric is a frequency count of total child communication acts.

OTHER OUTCOMES:
Change in Acceptability of Intervention Measure (AIM) | Measured weekly during baseline, intervention, and post-intervention. Through study completion, 3-4 months
  Informant-reported measure of the acceptability of an intervention and/or implementation strategy. This four item questionnaire is administered to determine the extent to which stakeholders believe an intervention (e.g., AAC intervention) or implementation strategy (e.g., training, coaching) is acceptable. This measure was designed to be pragmatic, and adapted to an intervention, organization, or population. This measure has substantive and discriminant content validity, structural validity (Cronbach's alpha = 0.85) and test-test reliability (Cronbach's alpha = 0.83). The metric is a total score with a range of 4 - 20. Higher scores indicate greater acceptability.
Change in Intervention Appropriateness Measure (IAM) | Measured weekly during baseline, intervention, and post-intervention. Through study completion, 3-4 months
  Informant-reported measure of the appropriateness of an intervention and/ or implementation strategy. This four item questionnaire is administered to determine the extent to which stakeholders believe an intervention (e.g., AAC intervention) or implementation strategy (e.g., training, coaching) is appropriate. The measure was designed to be pragmatic, and adapted to an intervention, organization, or population. This measure has substantive and discriminant content validity, structural validity (Cronbach's alpha = 0.91) and test-test reliability (Cronbach's alpha = 0.87). The metric is a total score with a range of 4 - 20. Higher scores indicate greater appropriateness.
Change in Feasibility of Intervention Measure (FIM) | Measured weekly during baseline, intervention, and post-intervention. Through study completion, 3-4 months
  Informant-reported measure of the feasibility of an intervention and/or implementation strategy. This four item questionnaire is administered to determine the extent to which stakeholders believe an intervention (e.g., AAC intervention) or implementation strategy (e.g., training, coaching) is feasible. The measure was designed to be pragmatic, and adapted to an intervention, organization, or population. This measure has substantive and discriminant content validity, structural validity (Cronbach's alpha = 0.89) and test-test reliability (Cronbach's alpha = 0.88). The metric is a total score with a range of 4 - 20. Higher scores indicate greater feasibility.
Change in Communication Complexity Scale (CCS; Aim 3 Only) | Study entry (start of study) and post-intervention (3-4 months later)
  Scripted assessment protocol with activities designed to elicit forms of communication. This assessment is used to describe the expressive communication skills of individuals who communicate using pre-symbolic and early symbolic behaviors. The CCS has adequate inter-observer agreement(k = 0.83), test-retest reliability ( r = 0.84), and concurrent validity with the Vineland II Expressive Communication Subscale (r = 0.47. The metric is the total optimal score with a range of 0 - 12. Higher scores indicate greater communication skills.
Change in Communication Matrix (Aim 3 Only) | Study entry (start of study) and post-intervention (3-4 months later)
  Assessment consisting of 24 questions to describe early expressive communication skills of individuals who primarily communicate using pre-symbolic and early symbolic behaviors. This Communication Matrix has high inter-rater reliability (0.96). The metric is a total score with a range of 0 - 160. Higher scores indicate greater communication skills.
Change in Preschool-Language Scales 5th Edition (Aim 3 Only) | Study Entry (start of study) and Post Intervention (3-4 months later)
  Standardized Assessment of expressive and receptive language skills. The metric is the total standard score with a mean of 100 and SD of 15

CONTACTS AND LOCATIONS:
Overall Officials: Emily D. Quinn, Ph.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
The final data set will include caregiver and SLP interview transcripts, standardized cognitive and language assessments, caregiver-reported demographic and behavioral data, observational data of the children in their caregivers at home over time and social validity questionnaires. This data set will be stripped of identifiers prior to release for sharing. We will make the data and associated documentation available to users only under a data-sharing agreement that provides for a commitment: (1) to use the data only for research purposes and not to identify any individual participant, (2) to secure the data using appropriate computer technology, (3) to destroy or return the data after analyses are completed, and (4) to cite the grant and key publications describing the database and measures in any resulting presentations and publications.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available one year after all of the data analysis is complete.
Access Criteria: We will make the data and associated documentation available to users only under a data-sharing agreement that provides for a commitment: (1) to use the data only for research purposes and not to identify any individual participant, (2) to secure the data using appropriate computer technology, (3) to destroy or return the data after analyses are completed, and (4) to cite the grant and key publications describing the database and measures in any resulting presentations and publications.